CLINICAL TRIAL: NCT03335293
Title: A Randomized Clinical Trial to Compare the Addition of Epinephrine (no Epinephrine, 100mcg, and 200mcg) to the Standard Dose of Hyperbaric Bupivacaine 12mg, Fentanyl 20mcg and Morphine 150mcg in Scheduled C-sections.
Brief Title: RCT of Epinephrine (None, 100mcg, and 200mcg) in a Hyperbaric Bupivacaine, Fentanyl and Morphine Spinal in C-sections.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to FDA constraints on the off label use of the medications we will not be able to conduct this evaluation.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB201702657 - A
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy; Cesarean Section
Keywords: pregnancy; repeat cesarean section; spinal anesthesia; bupivacaine; epinephrine; intrathecal; analgesia
MeSH Terms: conditions — Agnosia | interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): normal saline vehicle added to subarachnoid block
  Interventions: Other: normal saline
- 100 mcg epinephrine (Experimental): 100 mcg epinephrine added to subarachnoid block
  Interventions: Drug: 100 mcg Epinephrine
- 200 mcg epinephrine (Experimental): 200 mcg epinephrine added to subarachnoid block
  Interventions: Drug: 200 mcg Epinephrine

INTERVENTIONS:
Drug: 100 mcg Epinephrine — This study will evaluate the optimal dose of epinephrine as an adjunct to spinal doses of 1.6 mL hyperbaric bupivacaine + 20 mcg preservative free fentanyl + 150 mcg preservative-free morphine.
  Arms: 100 mcg epinephrine
Other: normal saline — placebo comparator
  Arms: Placebo
Drug: 200 mcg Epinephrine — This study will evaluate the optimal dose of epinephrine as an adjunct to spinal doses of 1.6 mL hyperbaric bupivacaine + 20 mcg preservative free fentanyl + 150 mcg preservative-free morphine.
  Arms: 200 mcg epinephrine

SUMMARY:
This is a prospective, randomized, double blind study of 75 patients (n=25 for each group) in which epinephrine (100mcg or 200mcg) or normal saline vehicle is added to intrathecal hyperbaric bupivacaine (0.75% bupivacaine hydrochloride in 8.25% dextrose), fentanyl, and morphine to prolong the duration of the spinal anesthetic in scheduled cesarean deliveries. The primary outcome of duration will be the time to T10 level sensory regression as well as motor level regression that will be graded via the modified Bromage scale.

Repeat cesarean sections, in particular, are associated with increased operative time and thus often performed with a spinal-epidural (CSE) technique. The epidural component is, however, untested and may not provide adequate anesthesia, thus the higher risk of conversion to a general anesthesia. Epinephrine is routinely used to prolong spinal anesthesia. If effective for the duration of a repeat cesarean section it would obviate the additional time and risks of performing the epidural and still avoid sufficient duration to avoid conversion to a general anesthetic.

DETAILED DESCRIPTION:
Spinal anesthesia is the most common type of anesthetic for C-section, but its major limitation is that the duration of the anesthesia may be less than the operative time. Repeat C-section is particularly associated with increased operative time and is often performed under a continuous spinal-epidural (CSE) technique. The epidural component is, however, untested and may not provide adequate anesthesia, thus necessitating the risk general anesthesia. Epinephrine may be used to prolong spinal anesthesia. This study will evaluate the optimal dose of epinephrine as an adjunct to usual spinal doses of 1.6 mL hyperbaric bupivacaine + 20 mcg preservative free fentanyl + 150 mcg preservative free morphine.

Adding epinephrine to hyperbaric bupivacaine helps in prolonging the duration of anesthesia and the quality of analgesia. However, the time to regression of the block effective for surgical anesthesia is not known for a C-section. Better quantification of this factor would help in choosing a spinal technique over a CSE in obstetric patients. This study seeks to quantify the duration of effective spinal anesthesia with the addition of either 100 or 200 mcg of epinephrine to an intrathecal mixture of hyperbaric bupivacaine and narcotics.

With early local anesthetics such as metycaine, nupercaine, or tetracaine, epinephrine was shown to intensify and prolonged their effects. Subsequent studies suggest that subarachnoid anesthesia with a combination of hyperbaric bupivacaine combined with an opioid and an adrenergic drug may be superior to techniques relying solely on local anesthetic drug. However, most of the studies were conducted in an orthopedic population for ambulatory and total joint arthroplasty for elderly patients.

Currently, it is well accepted that the addition of intrathecal narcotics will enhance the quality and duration of a spinal block.

Two investigations sought to determine the ED 95 dose of hyperbaric bupivacaine in combination with fentanyl and morphine to provide surgical anesthesia for operative success for cesarean delivery. Despite differences in spinal technique (sitting vs. lateral) the ED95 dose was 11.2 and 12 respectively. However, the mean duration of surgeries in those studies were significantly less (41 ± 15 and 64 ± 16 min respectively) than the mean duration of an elective C-section in our institution (90 ± 27 min with a 95th percentile of 135 min).

Since 12mg hyperbaric bupivacaine is the upper limit of acceptable doses for an elective C-section this study will evaluate the efficacy of epinephrine to extend the duration of effective surgical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective C-section patients
* ASA physical status class 1-3
* Age >18 years
* Height 140-180 cm
* Singleton pregnancy
* Gestational age ≥35 weeks

Exclusion Criteria:

* Age < 18 yo
* Prisoner status
* BMI > 45 Laboring patients with epidural going for emergency C-section Opioid abuse in the past 6 months Allergies to any of the adjuncts added to the spinal drug. Ruptured membranes four or more previous cesarean deliveries intrauterine growth retardation, abnormal placentation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
T4 sensory level | 15 minutes
  Time to T4 sensory level (this will be assessed by pin prick at the anterior axillary line)
T10 sensory regression | 120 minutes
  Time to regression to a T10 sensory level (this will be assessed by pinprick at the anterior axillary line)
Analgesia | 120 minutes
  Analgesia levels of the patient during the surgery (Pain scores will be measured at the beginning of surgery and during delivery, uterine manipulation, peritoneal suturing and skin closure. 0-10 pan scale)
Epidural dosing | 120 minutes
  Time elapsed after the spinal dose to the start of epidural dosing (this will be be assessed by review of the anesthesia record as the first recorded supplemental does of local anesthetic)
Satisfaction | 120 minutes and up to 24 hours after surgery
  Satisfaction levels of the patient during the surgery. (Maternal satisfaction will be quantified using a VAS score (0=no satisfaction and 100=full satisfaction) at the end of surgery and during a postoperative patient examination. )

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mongan, MD, Principal Investigator — UF COMJ Department of Anesthesiology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abouleish E, Rawal N, Fallon K, Hernandez D. Combined intrathecal morphine and bupivacaine for cesarean section. Anesth Analg. 1988 Apr;67(4):370-4. PMID 3354872
- [Background] Abouleish E, Rawal N, Rashad MN. The addition of 0.2 mg subarachnoid morphine to hyperbaric bupivacaine for cesarean delivery: a prospective study of 856 cases. Reg Anesth. 1991 May-Jun;16(3):137-40. PMID 1883770
- [Background] Abouleish E, Rawal N, Tobon-Randall B, Rivera-Weiss M, Meyer B, Wu A, Rashad MN. A clinical and laboratory study to compare the addition of 0.2 mg of morphine, 0.2 mg of epinephrine, or their combination to hyperbaric bupivacaine for spinal anesthesia in cesarean section. Anesth Analg. 1993 Sep;77(3):457-62. doi: 10.1213/00000539-199309000-00007. PMID 8368545
- [Background] Ginosar Y, Mirikatani E, Drover DR, Cohen SE, Riley ET. ED50 and ED95 of intrathecal hyperbaric bupivacaine coadministered with opioids for cesarean delivery. Anesthesiology. 2004 Mar;100(3):676-82. doi: 10.1097/00000542-200403000-00031. PMID 15108985
- [Background] Gurbet A, Turker G, Kose DO, Uckunkaya N. Intrathecal epinephrine in combined spinal-epidural analgesia for labor: dose-response relationship for epinephrine added to a local anesthetic-opioid combination. Int J Obstet Anesth. 2005 Apr;14(2):121-5. doi: 10.1016/j.ijoa.2004.12.002. PMID 15795147
- [Background] LEIMDORFER A, METZNER WR. Analgesia and anesthesia induced by epinephrine. Am J Physiol. 1949 Apr;157(1):116-21. doi: 10.1152/ajplegacy.1949.157.1.116. No abstract available. PMID 18144412
- [Background] Moore JM, Liu SS, Pollock JE, Neal JM, Knab JH. The effect of epinephrine on small-dose hyperbaric bupivacaine spinal anesthesia: clinical implications for ambulatory surgery. Anesth Analg. 1998 May;86(5):973-7. doi: 10.1097/00000539-199805000-00011. PMID 9585279
- [Background] Onishi E, Murakami M, Hashimoto K, Kaneko M. Optimal intrathecal hyperbaric bupivacaine dose with opioids for cesarean delivery: a prospective double-blinded randomized trial. Int J Obstet Anesth. 2017 May;31:68-73. doi: 10.1016/j.ijoa.2017.04.001. Epub 2017 Apr 13. PMID 28623089
- [Background] PRIDDLE HD, ANDROS GJ. Primary spinal anesthetic effects of epinephrine. Curr Res Anesth Analg. 1950 May-Jun;29(3):156-62. No abstract available. PMID 15414611